CLINICAL TRIAL: NCT03217422
Title: A Randomized, Double-blind, Placebo-controlled Study of the Safety and Efficacy of VAY736 in Autoimmune Hepatitis
Brief Title: ADCC Mediated B-Cell dEpletion and BAFF-R Blockade
Acronym: AMBER
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVAY736B2201; 2023-508859-39-00 (Registry Identifier: EU CT NUMBER)
Record Dates: First submitted 2017-07-12; First posted 2017-07-14 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Autoimmune Hepatitis
Keywords: Type 1; Type 2; autoimmune hepatitis; AIH
MeSH Terms: conditions — Hepatitis, Autoimmune | interventions — ianalumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind, placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1 (Experimental): VAY736 Dose 1
  Interventions: Biological: VAY736
- Arm 2 (Experimental): VAY736 Dose 2
  Interventions: Biological: VAY736
- Arm 3 (Experimental): VAY736 Dose 3
  Interventions: Biological: VAY736
- Arm 4 (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: VAY736 — VAY736
  Arms: Arm 1; Arm 2; Arm 3
Other: Placebo — Placebo control with conversion to active VAY736
  Arms: Arm 4

SUMMARY:
VAY736 dose testing; VAY736 efficacy and safety testing.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind dose range study in autoimmune hepatitis. The study population consists of female and male adult autoimmune hepatitis patients with incomplete response or intolerant to standard treatment of care. The diagnosis of autoimmune hepatitis has to fulfill the IAIHG criteria and must be confirmed by liver histology.

Patients will be randomly assigned to different doses of VAY736 or placebo. The primary analysis is planned at 24 weeks. A subsequent study part will then test the efficacy and safety of VAY736 in a parallel group design. For this part of the trial a new group of autoimmune hepatitis patients will be enrolled.

ELIGIBILITY:
Key Inclusion Criteria:

1. AIH diagnosed per International Autoimmune Hepatitis Group
2. Liver biopsy with Ishak modified HAI indicating active AIH
3. Incomplete response to OR intolerance of standard therapy (per AASLD)

Key Exclusion Criteria

1. Prior use of any B-cell depleting therapy (e.g., rituximab or other anti-CD20 mAb, anti-CD22 mAb or anti-CD52 mAb) within 1 year prior to Screening or as long as B-cell count <50 cells/µL
2. Required regular use of medications with known hepatotoxicity
3. Decompensated cirrhosis
4. Diagnosis of overlap syndrome with AIH (e.g., AIH+PBC, AIH+PSC).
5. Drug related AIH at screening or a history of drug related AIH.
6. History of drug abuse or unhealthy alcohol use
7. History of malignancy of any organ system
8. Pregnant or nursing (lactating) women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
ALT (Alanine aminotransferase) normalization | Week 24
  Difference in ALT normalization

SECONDARY OUTCOMES:
ALT normalization by dose | Week 24
  VAY736 dose-response

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Novartis Pharmaceuticals
Locations (27):
- United States (4):
  - Southern California Research Center, Coronado, California
  - Inland Empire Liver Foundation, Rialto, California
  - University of California Davis Medical Center, Sacramento, California
  - St. Lukes Advanced Liver Therapies, Houston, Texas
- Argentina (2):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, CABA
- Novartis Investigative Site, Ghent, Belgium
- Canada (3):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Novartis Investigative Site, Prague, Czechia
- Germany (5):
  - Novartis Investigative Site, Würzburg, Bavaria
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Mainz
- Japan (3):
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Takamatsu, Kagawa-ken
  - Novartis Investigative Site, Itabashi Ku, Tokyo
- Spain (2):
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Bern, Switzerland
- United Kingdom (5):
  - Novartis Investigative Site, Birmingham, West Midlands
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Newcastle upon Tyne
  - Novartis Investigative Site, Nottingham
  - Novartis Investigative Site, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Cholankeril G, Vierling JM. The clinical imperative of a complete biochemical response to immunosuppression in autoimmune hepatitis: Close is not good enough! Hepatology. 2024 Mar 1;79(3):529-531. doi: 10.1097/HEP.0000000000000597. Epub 2023 Sep 18. No abstract available. PMID 37722131
- [Derived] Chung YY, Rahim MN, Heneghan MA. Autoimmune hepatitis and pregnancy: considerations for the clinician. Expert Rev Clin Immunol. 2022 Apr;18(4):325-333. doi: 10.1080/1744666X.2022.2044307. Epub 2022 Mar 2. PMID 35179437